CLINICAL TRIAL: NCT04671875
Title: A Phase I Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of MIL93 in Advanced or Metastatic Solid Tumors.
Brief Title: A Clinical Study of MIL93 in Solid Tumors.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIL93-CT101
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-12

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIL93 (Experimental)
  Interventions: Drug: Recombinant Humanized Monoclonal Antibody MIL93

INTERVENTIONS:
Drug: Recombinant Humanized Monoclonal Antibody MIL93 — PART I :The patients confirming to the eligibility criteria will be assigned to the 6 dose groups (0.3mg/kg, 1mg/kg, 3mg/kg, 10mg/kg, 20mg/kg, 30mg/kg,respectively) based on the sequence of inclusion. Each patient will receive an intravenous infusion of MIL93 every 3 or 2 week on Day 1.
  PART II:One recommended dose will be conducted from 6 dose groups based on results of PART I.

SUMMARY:
MIL93 is a recombinant humanized anti-Claudin 18.2 (CLDN18.2) IgG1 monoclonal antibody. This is an open label Phase I study to evaluate safety, tolerability, pharmacokinetics and efficacy of MIL93 in Advanced or Metastatic solid tumors.

DETAILED DESCRIPTION:
This study is composed of two stages:Part I is mono-therapy dose escalation and dose expansion study, and Part II is the study of combination therapy.

The dose escalation study will be conducted using Part I for testing optimal doses at 0.3,1, 3, 10, 20, 30 mg/kg every 3 weeks (Q3W). An accelerated titration followed by traditional 3+3 design will be used in this study with a 21-day dose-limiting toxicity (DLT) observation period. Based on the data of dose escalation study, determine whether to carry out dose escalation at frequency of every 2 weeks(Q2W) and how many cohorts will be added in dose expansion study.

Based on the data of Part I, one or two doses will be conducted in the study of combination therapy. The study of PART II is composed of two cohorts. Cohort 1:Subjects with untreated CLDN18.2 positive gastric/gastroesophageal junction adenocarcinoma(G/GEJAC) will be treated with MIL93 and standard first-line chemotherapy.Cohort 2:Subjects with untreated CLDN18.2 positive pancreatic cancer will be treated with MIL93 and standard first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, >=18 years of age;
2. Suffer from advanced unresectable or metastatic malignant solid tumors confirmed by histological diagnosis and meet the criteria of the enrolled group as follows:

   Mono-therapy dose escalation study: The subjects for whom no standard treatment regimens are available or who is intolerable to standard treatments.

   Mono-therapy dose expansion study: The subjects with positive CDLN18.2 expression in tumor tissue (through immunohistochemistry (IHC) test) confirmed by the central laboratory at enrollment.

   Combination study is composed of 2 cohorts.Cohort 1:Subjects with untreated CLDN18.2 positive G/GEJAC; Cohort 2:Subjects with untreated CLDN18.2 positive pancreatic cancer.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. Life expectancy >=3 months;
5. Sufficient organ and bone marrow function;
6. At least one measurable lesion or evaluable lesion (recist v1.1);
7. Able and willing to provide written informed consent and to comply with the study protocol.

Exclusion Criteria:

1. Prior use of any anti-cancer therapy(including chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc) within 4 weeks of study start;
2. Previous exposure to any drug targeting CLDN 18.2;
3. Major surgery within 8 weeks prior to the first administration or expected to undergo major surgery during the study treatment;
4. Systemic immunosuppressive therapy was required within 14 days prior to the first administration;
5. Central nervous system metastasis;
6. History of other primary malignant tumors in 5 years;
7. Evidence of significant, uncontrolled concomitant disease;
8. Infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C(including HBsAg,HBcAb positive with abnormal HBV DNA or HCV RNA );
9. Suffering from serious or uncontrollable gastro-intestinal tract bleed;
10. Known severe allergic reaction or/and infusion reaction to monoclonal antibody;
11. Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) while participating in the study; 2) for at least 6 months after discontinuation of all study treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | up to 1year after enrollment
  Percentage of Participants with AEs and SAEs assessed by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Pharmacokinetics:AUC | up to 1year after enrollment
  The area under the curve (AUC) of serum concentration of the drug after the administration
Pharmacokinetics: Cmax | up to 1year after enrollment
  Maximum concentration(Cmax) of the drug after administration
Objective response rate (ORR) | up to 1year after enrollment
  To evaluate preliminary anti-tumor activity of MIL93 in subjects with advanced malignancies.ORR includes complete remission(CR) and partial remission(PR) assessed by RECIST v1.1 criteria.
Duration of response (DoR) | up to 1year after enrollment
  DOR is defined as the time from the initial response (CR or PR) to the time of disease progression or death, whichever occurs first.
Progression free survival (PFS) | up to 1year after enrollment
  Defined as the time from the first day of study treatment to disease progression or death, whichever occurs first.
Immunogenicity | up to 1year after enrollment
  Anti-Drug Antibodies (ADA) will be tested and percentage of ADA positive patients will be calculated to evaluate immunogenicity of MIL93.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China